CLINICAL TRIAL: NCT01230294
Title: Evaluation of New Echocardiographic Methods for Measurement of Right Ventricular Function.
Brief Title: New Echocardiographic Methods for Right Ventricular Function.
Acronym: NEW-RV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Derliz Mereles, Derliz Mereles, M.D., Heidelberg University
Other Study IDs: S275-2010
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Right Ventricular Dysfunction
Keywords: echocardiography of the right heart; 3D 4D echocardiography; strain measurement; chronic heart failure; pulmonary hypertension
MeSH Terms: conditions — Ventricular Dysfunction, Right; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- control: participants without structural heart disease
- CHF: patients with chronic heart failure of the left ventricle affecting the right heart
- PAH: patients with pulmonary arterial hypertension without left ventricular dysfunction

SUMMARY:
Aims of this study are the evaluation of new echocardiographic methods (3D/4D- and strain-echocardiography) for measurement of the right ventricular (RV) function .

DETAILED DESCRIPTION:
Studies of the last years revealed that the right ventricular function is an important predictive value for the survival of patients with congenital heart disease, pulmonary hypertension or chronic heart failure. In 2006 the National Heart, Lung and Blood Institute has pronounced the right ventricular dysfunction including the non-invasive assessment of the right ventricular function as preferential aim of cardiovascular research.

Many parameters are used to describe right ventricular dysfunction, but none of these has a comparable significance like the left ventricular ejection fraction. Because of the limitation of each right ventricular parameter the stepwise combination of these parameters is used to describe right ventricular function what frequently results in further problems, especially in comparison of long-term controls.

Aims of this study are the evaluation of new echocardiographic methods (3D/4D- and strain-echocardiography) for measurement of the right ventricular (RV) function. The study is carried out as prospective, monocentric trial at the Department of Cardiology of the University Hospital of Heidelberg. Three different groups are set up for the assessment of the right ventricular function: patients with pulmonary arterial hypertension, patients with chronic heart failure of the left ventricle affecting the right heart and patients without structural heart disease who underwent an echocardiographic examination for other reasons (control group).

All participants are re-examined in constant intervals as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* persons of 18 years and older who receive a transthoracic echocardiography at our department
* written consent

Exclusion Criteria:

* present atrial fibrillation/flutter
* permanent pacemaker rhythm
* moderate/severe valvular heart disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * patients with pulmonary aterial hypertension
  * patients with chronic heart failure of the left ventricle affecting the right heart
  * patients without structural heart disease who underwent an echocardiographic examination for other reasons (control group)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
3D-volumetry of the right ventricle | 2 years
2D strain of the right ventricle | 2 years

SECONDARY OUTCOMES:
pulmonary artery systolic pressure (PASP) | 2 years
  standard value: ≤ 30 mmHg
tricuspid annular plane systolic excursion (TAPSE) | 2 years
  standard value: ≥ 20 mm
tricuspid annular systolic velocity (TASV) | 2 years
  standard value: ≥ 20cm/s
Tei-index (myocardial performance index) | 2 years
  standard value: ≥ 0,5
LV-eccentricity-index (Lei-index) | 2 years
  standard value: ≥ 1,0

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Greiner, M.D., Principal Investigator — Heidelberg University; Derliz Mereles, M.D., Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Greiner S, Andre F, Heimisch M, Hess A, Steen H, Katus HA, Mereles D. Non-invasive quantification of right ventricular systolic function by echocardiography: a new semi-automated approach. Clin Res Cardiol. 2013 Mar;102(3):229-35. doi: 10.1007/s00392-012-0528-z. Epub 2012 Dec 4. PMID 23208080
- [Derived] Greiner S, Goppelt F, Aurich M, Katus HA, Mereles D. Prognostic relevance of the right ventricular myo-mechanical index (RV-MMI) in patients with precapillary pulmonary hypertension. Open Heart. 2018 Sep 12;5(2):e000903. doi: 10.1136/openhrt-2018-000903. eCollection 2018. PMID 30245839
- [Derived] Greiner S, Heimisch M, Aurich M, Hess JA, Katus HA, Mereles D. Multiplane two-dimensional strain echocardiography for segmental analysis of right ventricular mechanics: new-RV study. Clin Res Cardiol. 2014 Oct;103(10):817-24. doi: 10.1007/s00392-014-0723-1. Epub 2014 May 16. PMID 24830514